CLINICAL TRIAL: NCT06224114
Title: A Pilot, Randomised, Masked Study to Investigate the Effect of Coloured-light on Colour Contrast Thresholds in Retinitis Pigmentosa.
Brief Title: Coloured-light in Retinitis Pigmentosa.
Acronym: CLIRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 161090
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Inherited eye disease; Retinal dystrophy; Retinitis Pigmentosa; Visual impairment; Photobiomodulation; Mitochondrial Dysfunction
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Dystrophies; Vision Disorders; Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Technicians responsible for study measurements, Chief Investigator (CI), Principal Investigator (PI) and collaborators will be masked to the treatment allocation. It is not possible for participants to be fully masked as they will know which wavelength (colour) of light they have been provided, but they will not be told which wavelength of light is the active intervention. Participants will be advised not to discuss the colour of light used with the masked technicians and study team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coloured light 1 group (Experimental): Coloured light 1 group will be provided with a coloured-light torch and instructed to apply it to their study eye for 3 minutes at home each morning between 8 - 10 am for 28 days.
  Interventions: Device: Coloured-light torch
- Coloured light 2 group (Placebo Comparator): Coloured light 2 group will be provided with a different coloured-light torch and instructed to apply it to their study eye for 3 minutes at home each morning between 8 - 10 am for 28 days.
  Interventions: Device: Different coloured-light torch

INTERVENTIONS:
Device: Coloured-light torch — Participant administered, at-home, 3-minute daily morning application (between 8 - 10am) of a coloured-light torch to the study eye.
  Arms: Coloured light 1 group
Device: Different coloured-light torch — Participant administered, at-home, 3-minute daily morning application (between 8 - 10am) of a different coloured-light torch to the study eye.
  Arms: Coloured light 2 group

SUMMARY:
This study will assess the effect of 2 different colours of light on colour vision in adults with retinitis pigments (RP). Participants will be 18 years or above with a genetically confirmed molecular diagnosis of RP. After informed consent, participants will have their letter chart vision and colour vision measured in their study eye. They will then be they will be randomly allocated to one of 2 groups. The study team will not know which group they have been assigned to. Group 1 will be given a coloured-light hand-held torch and be asked to apply it to their study eye for 3 minutes at home each morning between 8 - 10 am for 28 days. Group 2 will be given a different colour hand-held torch and be asked to do the same. All participants will have their letter chart vision and colour vision measured at the end of study on day 28 (+ 7 days).

DETAILED DESCRIPTION:
This is a pilot, randomised, masked, single-site trial designed to assess the effect of coloured light exposure on cone contrast thresholds (CCT) in adults with RP.

70 adults with typical RP in which the underlying genetic cause is known will be recruited from Moorfields Eye Hospital genetics service.

Following informed consent, participants will be invited for a baseline study visit.

At a baseline visit, prior to any light exposure (day 0), participants will undergo Logarithm of the Minimum Angle of Resolution (LogMAR) visual acuity (VA) and CCT measurements performed by an experienced technician according to dedicated standard operating procedures. The order of testing will be as follows:

* Study eye: LogMAR VA
* Study eye: CCT (Tritan and Protan)

After baseline assessments have been completed, participants will be randomised to the intervention (n=35) or control group (n=35) by a study nurse. All other study team members will be masked to group allocation.

The intervention group will be provided with a coloured torch and instructed to apply it to their study eye for 3 minutes at home each morning between 8 - 10 am for 28 days. The control group will be provided with a different coloured torch and will be instructed to follow the same protocol. The specific colours have not be disclosed here to protect masking of the study. Participants will be asked to complete a paper diary each day to record whether light was applied, the time and duration of the application and the eye to which light was applied.

The end of trial visit will be scheduled on day 28 (+7 days). Participants will undergo LogMAR VA and CCT measurements by an experienced technician according to standard operating procedures (SOP). The order of testing will be as follows:

* Study eye: LogMAR VA
* Study eye: CCT (Tritan and Protan)

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Typical RP where the underlying genetic cause is known. This may include PRPF31, PRPF8, SNRNP200, RHO, RP1 [autosomal dominant] and USH2A, EYS [autosomal recessive]
* VA of 0.30 LogMAR (6/12) or better in the study eye
* Preserved foveal structure defined by intact outer retinal (ellipsoid zone) at the fovea on Optical Coherence Tomography (OCT) and a hyperfluorescent ring within the temporal vascular arcades on Fundus Autofluorescence (FAF) in the study eye
* Willing and able to provide written informed consent

Exclusion Criteria:

* Co-existing ocular pathology will be excluded; however, participants with macular oedema, a common pre-symptomatic manifestation of foveal involvement, will not be excluded
* Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within 6 months of study enrolment
* Unwilling or able to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Tritan Colour Contrast Threshold (CCT) | Measured at Day 0 and Day 28
  Tritan CCT will be measured using the ChromaTest® platform, a software program which quantifies age-corrected tritan and protan CCT using a Modified Binary Search method. Tritan CCT test endpoint is a continuous variable (units: percentage).

SECONDARY OUTCOMES:
Protan CCT | Measured at Day 0 and Day 28
  Protan CCT will be measured using the ChromaTest® platform, a software program which quantifies age-corrected tritan and protan CCT using a Modified Binary Search method. Protan CCT test endpoint is a continuous variable (units: percentage).
LogMAR Visual Acuity (LogMAR VA) | Measured at Day 0 and Day 28
  LogMAR VA will be measured on an electronic LogMAR acuity chart (Test Chart 2020, Thompson Software Solutions, UK), according to a forced-choice procedure.
Proportion of participants losing ≥15 letters of LogMAR VA | Measured each day (Day 0 through Day 28)
  Proportion of participants losing 15 letters of LogMAR VA or more at day 28 will be reported as a safety outcome.
Compliance rate | Measured each day (Day 0 through Day 28)
  Compliance rate of application of daily, 3-minute, at-home, participant administered coloured-light exposure is a secondary endpoint. This will be collected through completion of a participant diary.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Dunbar, PhD, Principal Investigator — UCL Institute of Ophthalmology
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers